CLINICAL TRIAL: NCT03652090
Title: Evaluation of the Primary Human Nasal Epithelial Cell Culture Model in the Context of Personalized Therapy in Cystic Fibrosis
Brief Title: Primary Nasal Cell Culture as a Tool for Personalized Therapy in Cystic Fibrosis
Acronym: Epiithelix
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: ABCF2 (Unknown)
Responsible Party: Principal Investigator, Isabelle Sermet-Gaudelus, Professor, Institut National de la Santé Et de la Recherche Médicale, France
Other Study IDs: 2010-05-03 A3
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
Keywords: biomarker
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — p
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- cystic fibrosis patients: Cystic fibrosis patients carrying to 2 CFTR mutations undergoing cell sampling
  Interventions: Procedure: cell sampling
- healthy heterozygotes: healthy heterozygotes carrying 1 CFTR mutations undergoing cell sampling
  Interventions: Procedure: cell sampling
- healthy control: subject with no evidence of any symptoms compatible with Cystic Fibrosis undergoing cell sampling
  Interventions: Procedure: cell sampling

INTERVENTIONS:
Procedure: cell sampling — nasal brushing to collect cells

SUMMARY:
characterization of CFTR function and expression in nasal primary cells collected from patients with cystic fibrosis in comparison to their parents, healthy heterozygotes and healthy controls

DETAILED DESCRIPTION:
3 groups of subjects are enrolled CF subjects according to their genotypes (aiming to enroll patients carrying 2 CF causing mutations with no CFTR expression/function, and patients carrying at least 1 mutation with residual function, such R117H) Parents or siblings of the CF subjects, as healthy hétérozygotes healthy controls All these subjects experience nasal brushings. From these nasal brushings,nasal cells are expanded, and cultured in air liquid interface to obtain polarized epithelium. This epithelium is then studied in Ussing chamber experiments to characterize the level of cAMP dependant Chloride transport and Sodium reabsorption. Apical expression of CFTR is assessed by immunofluorescence.

Results will allow to define the variability of CFTR function and expression criteria in subjects with the same genotype. Such data are crucial for interpretation of the effect of CFTR modulators.

ELIGIBILITY:
Inclusion Criteria:

* patients with Cystic Fibrosis with 2 mutations in CFTR
* healthy heterozygotes with 1 mutation in CFTR
* healthy subjects with no familial history of Cystic Fibrosis and no symptoms suggesting Cystic Fibrosis

Exclusion Criteria:

* smoking

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with Cystic Fibrosis with 2 mutations in CFTR
  * healthy heterozygotes with 1 mutation in CFTR
  * healthy subjects with no familial history of Cystic Fibrosis and no symptoms compatibel with Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
variation in the short-circuit-current (Isc) after Forskolin (Forskolin)/IBMx and VX-770 (∆IscFsk/IBMx+VX-770) | 1 day
  The short-circuit-current (Isc) was measured under voltage clamp conditions. Inhibitors and activators were added after stabilization of baseline Isc. The sum of the change after Forskolin (Forskolin)/IBMx and VX-770 (∆IscFsk/IBMx+VX-770) served as an index of CFTR function.

SECONDARY OUTCOMES:
percentage of cells displaying apical staining | 1 day
  CFTR immuno-detection was performed as previously described 31. Apical CFTR staining was assessed semi quantitatively as the percentage of cells displaying apical staining multiplied by the average corrected apical fluorescence 32.